CLINICAL TRIAL: NCT03096405
Title: Impact MRSA -PCR on Patient Management
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: PCR-SARM
Record Dates: First submitted 2017-03-25; First posted 2017-03-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-03

CONDITIONS: MRSA Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Polymerase Chain Reaction of Methicillin Resistant Staphyloccus Aureus — Polymerase Chain Reaction of Methicillin Resistant Staphyloccus Aureus

SUMMARY:
Staphylococcus aureus represents one of the most met germs, with Escherichia coli, during bacteremia. Microbiologist distinguish at aureus S. two profiles of resistance in beta-lactamines: S. aureus sensitive to the methicillin ( SASM) and the S. aureus resistant to the methicillin ( SARM).

With the implementation of the MALDI-TOF, it is now possible to identify the origin responsible of the bacteremia the day of the positivity of the hemoculture ( J0) and to set up a treatment with adapted antibiotic, which, in the case of a sepsis to aureus S., is the vancomycine. Ye it was demonstrated, that the use of the vancomycine on the SASM increased the average duration of stay and a more important rate of relapse.

The PCR SARM was organized in the GHPSJ in 2014. It allows from the day of the positivity of the hemoculture ( J0), to determine the phenotype of resistance of S. aureus.

ELIGIBILITY:
Inclusion Criteria:

* Hemoculture positive to Staphylococcus Aureus Methicillin Sensitive

Exclusion Criteria:

* Positive test to Staphylococcus Aureus Methicillin Sensitive but not hospitalized.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: every patient hospitalized in St Joseph Hospital with an positive hemoculture to Staphylococcus Aureus Methicillin Sensitive
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Adaptation duration of antibiotherapy | 24 hours

SECONDARY OUTCOMES:
Mortality | Day 30
average duration of hospitalization | day 30

CONTACTS AND LOCATIONS:
Overall Officials: MIZRAHI Assaf, MD, Principal Investigator — Groupe Hospitalier Paris St JOSEPH; LEMONNIER Alban, MD, Study Chair — Groupe Hospitalier Paris St JOSEPH
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No